CLINICAL TRIAL: NCT01310569
Title: Relationship of Subcutaneous Adipose Tissue With HOMA-IR and Plasma Adiponectin Levels in Cases With Polycystic Ovarian Syndrome
Brief Title: Subcutaneous Adipose Tissue in Cases With Polycystic Ovarian Syndrome
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Aydogan Aydogdu, Gulhane School of Medicine
Other Study IDs: 27.04.2010/1491-764-10
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2010-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS, Skinfold thickness, HOMA-IR
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aimed to search whether whole body and subcutaneous adipose tissues increase in PCOS patients and whether these tissues are related to HOMA-IR and plasma adiponectin levels.

DETAILED DESCRIPTION:
Fifty-two patients with PCOS and fifty-tree healthy controls who were matched for body mass index (BMI) and age (p=0.430, p=0.112, respectively) were enrolled in the study. Biceps, triceps, subscapular and suprailiac skinfold thicknesses (SFT) of all cases were measured via caliper device; mid-upper arm circumference (MUAC) via a tape; and body fat distributions via a bioelectrical impedance device. Insulin resistance was calculated via HOMA-IR while ELISA was used to measure plasma adiponectin.

ELIGIBILITY:
Inclusion Criteria:

* All of the women with PCOS had normal thyroid-stimulating hormone and prolactin (PRL) levels.

Exclusion Criteria:

* Subjects with possible ovarian tumors, congenital adrenal hyperplasia, BMI greater than 35 kg/m2, any chronic renal or liver disease, were excluded from the study.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with PCOS witout any other metabolik diseases
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Relationship of Subcutaneous Adipose Tissue with HOMA-IR and Plasma Adiponectin Levels in Cases with Polycystic Ovarian Syndrome | 2 year
  PCOS patients (the experimental group) had higher mean SFT values in all parts, mid-upper arm circumference values, whole body and trunk fat free mass amounts (FFM) and HOMA-IR values, while a lower adiponectin level.

CONTACTS AND LOCATIONS:
Overall Officials: Aydogan Aydogdu, MD, Study Director — Gulhane School of Medicine
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)